CLINICAL TRIAL: NCT00573768
Title: A Randomized, Double-blind, Multi-center, Vehicle-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Diclofenac Diethylamine 2.32% Gel Applied Once or Twice Daily in Patients With Acute Ankle Sprain
Brief Title: Efficacy and Safety of Diclofenac Diethylamine 2.32% Gel in Patients With Acute Ankle Sprain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VOPO-PE-201
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2010-10

CONDITIONS: Ankle Sprain
Keywords: Ankle, sprain, diclofenac diethylamine
MeSH Terms: conditions — Ankle Injuries; Sprains and Strains | interventions — diclofenac diethylamine; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: Diclofenac diethylamine 2.32% gel
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 3 (Active Comparator)
  Interventions: Drug: Diclofenac diethylamine 2.32% gel / Placebo

INTERVENTIONS:
Drug: Diclofenac diethylamine 2.32% gel — Diclofenac diethylamine 2.32% gel twice daily
  Arms: 1
Drug: Placebo — Vehicle 2 times daily
  Arms: 2
Drug: Diclofenac diethylamine 2.32% gel / Placebo — Diclofenac diethylamine 2.32% gel once daily / Vehicle once daily
  Arms: 3

SUMMARY:
This study will evaluate the efficacy of diclofenac diethylamine 2.32% gel in the treatment of acute ankle sprain.

ELIGIBILITY:
Inclusion Criteria:

* Acute sprain of the ankle
* Injury within past 48 hours.

Exclusion Criteria:

* Pain medication taken since the injury
* Pain or instability in the same ankle due to previous ankle sprain or any other trauma.
* Ankle sprain due to a known disease affecting the ligaments

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2007-11; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Baltzer, Principal Investigator
Locations (21):
- Germany (21):
  - Novartis Investigative Site, Bad Bramstedt
  - Novartis Investigative Site, Bad Nauheim
  - Novartis Investigative Site, Bad Zwischenahn
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Eichstätt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hammelburg
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Kaufbeuren
  - Novartis Investigative Site, Lambrecht/Pfalz
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Meersburg
  - Novartis Investigative Site, Munich
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neustadt/Aisch
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Stockach

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start 27 Nov 2007 Recruitment end 26 Jun 2007 Private Practices
Groups:
- Diclofenac Diethylamine (DDEA) 2.32% Gel BID: Twice daily (BID) application
- DDEA 2.32% Gel OD: Once daily (OD) application of active gel and OD application of vehicle gel
- Vehicle Gel: BID application
Period: Overall Study
Arm/Group | Diclofenac Diethylamine (DDEA) 2.32% Gel BID | DDEA 2.32% Gel OD | Vehicle Gel
Started | 89 | 91 | 91
Completed | 87 | 89 | 87
Not Completed | 2 | 2 | 4
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Diethylamine (DDEA) 2.32% Gel BID | DDEA 2.32% Gel OD | Vehicle Gel | Total
Number analyzed (Participants) | 89 | 91 | 91 | 271
Age Continuous [Mean (Standard Deviation); unit: years] | 38.8 (13.7) | 38.2 (14.6) | 38.9 (14.1) | 38.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 47 | 46 | 142
  Male | 40 | 44 | 45 | 129
Region of Enrollment [Number; unit: participants]
  Germany | 89 | 91 | 91 | 271

OUTCOME MEASURES:

1. Primary Outcome: Pain on Movement on Day 5 (Change From Baseline). A Greater Change From Baseline on Day 5 Equates to a Better Outcome.
Description: Pain on movement: visual analogue scale (VAS) with anchors at 0 mm (no pain) and 100 mm (extreme pain)
Time Frame: change from baseline (on day 1) to day 5
Population: Intent to treat (ITT)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac Diethylamine (DDEA) 2.32% Gel BID | DDEA 2.32% Gel OD | Vehicle Gel
Number analyzed (Participants) | 89 | 91 | 91
mm | 38.3 (22.7) | 35.7 (20.4) | 33.4 (20.9)

ADVERSE EVENTS:
Arm/Group | Diclofenac Diethylamine (DDEA) 2.32% Gel BID | DDEA 2.32% Gel OD | Vehicle Gel
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/91 | 0/91
Other Adverse Events (participants affected / at risk) | 3/89 | 6/91 | 1/91
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diclofenac Diethylamine (DDEA) 2.32% Gel BID (N=89) | DDEA 2.32% Gel OD (N=91) | Vehicle Gel (N=91)
headache (Nervous system disorders) | 3 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No